CLINICAL TRIAL: NCT01363999
Title: A Single-center, Randomized, Open-label, Four Treatments, Four Periods, Four Sequence, Four-way Crossover Study to Explore the Pharmacokinetic Performance of Dalcetrapib and Atorvastatin Fixed Dose Combination Prototype Formulations in Healthy Volunteers
Brief Title: A Formulation Screening Study of Dalcetrapib and Atorvastatin in Healthy Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: WP25642
Record Dates: First submitted 2011-05-31; First posted 2011-06-02 (Estimated); Results first posted 2019-12-17 (Actual); Last update posted 2019-12-17 (Actual); Status verified 2019-12

CONDITIONS: Healthy Volunteer
MeSH Terms: interventions — Atorvastatin; dalcetrapib

ARMS (4):
- A (Experimental): RO5317116/F01 bilayer tablet
  Interventions: Drug: atorvastatin; Drug: dalcetrapib
- B (Experimental): RO5317116/F03 bilayer tablet
  Interventions: Drug: atorvastatin; Drug: dalcetrapib
- C (Experimental): RO5317116/F04 active-coated tablet
  Interventions: Drug: atorvastatin; Drug: dalcetrapib
- D (Experimental): RO4607381/F49 tablet
  Interventions: Drug: atorvastatin; Drug: dalcetrapib

INTERVENTIONS:
Drug: atorvastatin — single dose of atorvastatin on day 1
Drug: dalcetrapib — single dose of dalcetrapib on day 1

SUMMARY:
A single-center, crossover study to evaluate the pharmacokinetics of dalcetrapib and atorvastatin from prototype fixed dose combination formulations in healthy volunteers. Volunteers will receive a single dose of dalcetrapib with atorvastatin in each of four treatment periods.

ELIGIBILITY:
Inclusion Criteria:

* Healthy volunteers, 18 to 55 years of age, inclusive

Exclusion Criteria:

* Any concomitant disease or ongoing condition that in the investigator's opinion could interfere with the study or could pose an unacceptable risk to the patient
* Clinically significant abnormal laboratory values

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 24 (Actual)
Dates: Start 2011-06; Primary Completion 2011-07 (Actual); Study Completion 2011-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (1):
- Christchurch, New Zealand

RESULTS

PARTICIPANT FLOW:
Groups:
- Total Study: All AE and Demographic Data is listed for the Total Study Population
Period: A: RO5317116/F01 Bilayer Tablet
Arm/Group | Total Study
Started | 24
Completed | 24
Not Completed | 0
Period: B: RO5317116/F03 Bilayer Tablet
Arm/Group | Total Study
Started | 24
Completed | 24
Not Completed | 0
Period: C: RO5317116/ F04 Active-coated Tablet
Arm/Group | Total Study
Started | 24
Completed | 24
Not Completed | 0
Period: D: RO4607381/ F49 Tablet
Arm/Group | Total Study
Started | 24
Completed | 24
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Total Study
Number analyzed (Participants) | 24
Age, Continuous [Mean (Standard Deviation); unit: years] | 27.1 (9.77)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 15
  Male | 9

OUTCOME MEASURES:

1. Primary Outcome: Plasma Concentration of Dalcetrapib Active Form
Time Frame: 3 days
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Groups:
- A, RO5317116/F01 Bilayer Tablet: RO5317116/F01 bilayer tablet
  atorvastatin: single dose of atorvastatin on day 1
  dalcetrapib: single dose of dalcetrapib on day 1
- B, RO5317116/F03 Bilayer Tablet: RO5317116/F03 bilayer tablet
  atorvastatin: single dose of atorvastatin on day 1
  dalcetrapib: single dose of dalcetrapib on day 1
- C, RO5317116/F04 Active-coated Tablet: RO5317116/F04 active-coated tablet
  atorvastatin: single dose of atorvastatin on day 1
  dalcetrapib: single dose of dalcetrapib on day 1
- D, RO4607381/F49 Tablet: RO4607381/F49 tablet
  atorvastatin: single dose of atorvastatin on day 1
  dalcetrapib: single dose of dalcetrapib on day 1
Arm/Group | A, RO5317116/F01 Bilayer Tablet | B, RO5317116/F03 Bilayer Tablet | C, RO5317116/F04 Active-coated Tablet | D, RO4607381/F49 Tablet
Number analyzed (Participants) | 24 | 24 | 24 | 24
ng/mL | 285 (68.2) | 272 (61.9) | 294 (42) | 231 (55.9)

2. Primary Outcome: Plasma Concentration of Atorvastatin
Time Frame: 3 days
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | A, RO5317116/F01 Bilayer Tablet | B, RO5317116/F03 Bilayer Tablet | C, RO5317116/F04 Active-coated Tablet | D, RO4607381/F49 Tablet
Number analyzed (Participants) | 24 | 24 | 24 | 24
ng/mL | 3.56 (46.5) | 3.55 (50.8) | 4.26 (60.8) | 3.86 (61.2)

3. Secondary Outcome: Plasma Concentration of Atorvastatin Metabolites
Description: Measuring the amount of byproducts of the metabolization of Atorvastatin in the blood plasma.
Time Frame: 3 days
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/ml
Arm/Group | A, RO5317116/F01 Bilayer Tablet | B, RO5317116/F03 Bilayer Tablet | C, RO5317116/F04 Active-coated Tablet | D, RO4607381/F49 Tablet
Number analyzed (Participants) | 24 | 24 | 24 | 24
ng/ml | 2.50 (37.2) | 2.51 (50.7) | 2.95 (46.9) | 2.77 (51.5)

4. Secondary Outcome: Safety: Incidence of Serious Adverse Events
Time Frame: 9 weeks
Measure: Number; unit: Events
Arm/Group | A, RO5317116/F01 Bilayer Tablet | B, RO5317116/F03 Bilayer Tablet | C, RO5317116/F04 Active-coated Tablet | D, RO4607381/F49 Tablet
Number analyzed (Participants) | 24 | 24 | 24 | 24
Events | 0 | 0 | 0 | 0

ADVERSE EVENTS:
Groups:
- Total Study: All AE and Demographic Data is listed for the Total Study Population. Data was not collected by arm since all interventions contained the same formulation.
Arm/Group | Total Study
Serious Adverse Events (participants affected / at risk) | 0/24
Other Adverse Events (participants affected / at risk) | 8/24
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Total Study (N=24)
Appendectomy (Surgical and medical procedures) | 2
Inguinal Hernia Repair (Surgical and medical procedures) | 2
Seasonal Allergy (Immune system disorders) | 4

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No